CLINICAL TRIAL: NCT02039973
Title: Healthy Options: Group Psychotherapy for HIV-positive Depressed Perinatal Women.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Harvard Medical School (HMS and HSDM) (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Mary Kay Smith Fawzi, Assistant Professor of Global Health and Social Medicine, Harvard Medical School (HMS and HSDM)
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: 1R01MH100338-01 (NIH); 1R01MH100338-01 (NIH)
Record Dates: First submitted 2014-01-01; First posted 2014-01-20 (Estimated); Last update posted 2018-02-22 (Actual); Status verified 2018-02

CONDITIONS: Depression
Keywords: HIV; AIDS; Tanzania; depression; perinatal; psychotherapy; task-sharing; problem-solving
MeSH Terms: conditions — Depression; Acquired Immunodeficiency Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Task-sharing approach to group therapy (Experimental): The intervention will consist of problem-solving therapy as well as cognitive behavioral components. Core problem-solving therapy components will involve lay CBHW facilitated discussions to explore symptoms of depression and how problems are related to depression. Core cognitive behavioral components will include lay CBHW facilitated discussions to explain the purpose of the sessions, as well as effect a number of behavioral changes in participants.
  Interventions: Behavioral: Task-sharing approach to group therapy
- Enhanced standard of care (Active Comparator): The control condition will promote an enhanced standard of care. Clinicians and nurses at MCH clinics included in the study will receive a structured one day re-orientation training consistent with the World Health Organization (WHO) mh-GAP guidelines for assessment as well as basic psychosocial and drug treatment of moderate to severe depression in primary care settings. The training will be consistent with the standard of care for mental health among HIV-positive populations as outlined in Tanzanian health policy. In addition, clinical staff will be trained to encourage women to invite their male partners to accompany them at clinic visits, where psycho-education on perinatal depression for couples will be offered for those opting to participate.
  Interventions: Behavioral: Enhanced standard of care

INTERVENTIONS:
Behavioral: Task-sharing approach to group therapy — Participants will also identify, select and clarify common concerns/problems; provide orientation to steps in problem-solving; break down identified problems into manageable pieces; choose pieces of problem to address in facilitated discussion of problem solving for implementing solutions; support the sharing of feedback of strategies used in problem-solving and maintaining pleasurable activities.
  Additionally, the intervention to aim to effect behavior by: explaining the links between problems, negative thoughts, choices made on a day-to-day basis, behaviors, and mood (symptoms of depression); facilitate sharing of practical skills to tackle problems, to change mood-related thoughts, choices and/or behaviors; offer and provide feedback on homework assignments to encourage practice of skills; and help participants attribute reported improvements to the use of new skills during feedback sessions.
  Arms: Task-sharing approach to group therapy
Behavioral: Enhanced standard of care
  Arms: Enhanced standard of care

SUMMARY:
Although there is a significant burden of depression among HIV-positive women in Tanzania, there is a critical gap between the needs of this population and the integration of mental health and PMTCT-plus services. The long-term intent of the research is to bridge this gap with the overall goal to examine the potential for successful integration of enhanced mental health care and brief group interventions among HIV-positive women receiving PMTCT-plus services and to evaluate a combination of evidence-based approaches for treatment of depression in this vulnerable population in Tanzania.

DETAILED DESCRIPTION:
In resource-limited settings, there has been a significant increase in access to antiretroviral therapy (ART) in recent years. Although there remain serious limitations in access to ART in these settings, for many who have initiated and continue treatment, HIV disease is a chronic condition that needs to be managed over time. There is considerable evidence that individuals with chronic illness have an increased risk of depression, in part related to the challenges in coping and managing their illness. Rates for depression during pregnancy in women living with HIV are estimated to be higher.

Despite this relatively high burden of depression among persons living with HIV/AIDS (PLHA), it has been documented that clinical staff working with PLHA do not routinely identify or treat depression in this setting. This is in contrast to recent revisions in the Tanzanian health policy that emphasize integrating mental health and HIV care at district and lower level health care services. The long-term intent of the research is to bridge this gap between Tanzanian health policy and implementation of integrating mental health care among pre- and post-natal women receiving HIV care. Therefore, the overall goal of the proposed study is to examine the potential for successful integration of enhanced mental health care and group counseling among HIV-positive women receiving preventing mother to child transmission (PMTCT)-plus services and to evaluate a combination of evidence-based approaches in treatment of depression in this vulnerable population in Tanzania.

Specifically this application aims to:

1. Examine the acceptability and feasibility of integrating an enhanced standard of mental health care and group counseling with PMTCT-plus services provided at government-run maternal and child health (MCH) clinics, from the perspectives of: a) facility mental health care focal points and MCH clinic managers, b) perinatal direct care providers; and c) HIV-positive perinatal women;
2. Validate a depression screening tool for major depressive disorder (MDD) and suicidality for use in Tanzania; and
3. Conduct a cluster randomized controlled trial comparing a task-sharing approach (i.e. problem solving and cognitive behavioral therapy components delivered to groups facilitated by lay community based health care workers (CBHWs) versus improved standard

ELIGIBILITY:
Inclusion Criteria:

* pregnant women who access PMTCT-plus services at MCH clinics in Dar es Salaam
* HIV-positive serostatus
* screen positive for depression
* less than 28 weeks of gestation
* confirm they will attend postnatal services at the maternal and child health service they enrolled in for antenatal care for at least two years after they give birth

Exclusion Criteria:

* any woman less than 18 years of age
* HIV-negative
* screened negative for depression
* screened positive for depression and assessed to be of high suicide risk requiring immediate emergency referral for care
* not able to continue to receive care at the MCH clinic where they were initially enrolled for at least two years after giving birth

Ages: 18 Years to 49 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 742 (Actual)
Dates: Start 2013-07-01 (Actual); Primary Completion 2017-12-31 (Actual); Study Completion 2017-12-31 (Actual)

PRIMARY OUTCOMES:
Depressive disorder and suicidality | Q3 2016 after an average of 1.5 years of follow-up
  Using a cut-off score based on the validation study, participants will be classified as having depressive and or suicidality or not. The trial aims to reduce rates of depression and suicidality among participants.

SECONDARY OUTCOMES:
Social support | Q3 2016 after an average of 1.5 years of follow-up
  For this measure, the Duke University-University of North Carolina Functional Social Support Questionnaire will be used; this scale has demonstrated positive correlations with other social support scales. A listing of ten items from this of this questionnaire has been used previously in Tanzania, reflecting dimensions of instrumental and emotional support
Self-Efficacy | Q3 2016 after an average of 1.5 years of follow-up
  The General Self-Efficacy Scale will be used to assess self-efficacy. This scale has demonstrated good internal consistency (Cronbach's alpha ranging from 0.81 to 0.91) and construct validity was shown through positive correlations with optimism and negative correlations with depression and anxiety.
HIV-related stigma | Q3 2016 after an average of 1.5 years of follow-up
  The HIV Stigma Scale developed by Berger et al. will be used to assess stigma; it has been validated in a diverse sample in the U.S. demonstrated construct validity through factor analysis and internal consistency (Cronbach's alpha of 0.96). A sub-sample of these items also demonstrated construct validity of this scale has also been demonstrated in a resource-limited setting.
Intimate partner violence | Q3 2016 after an average of 1.5 years of follow-up
  For intimate partner violence (IPV) the WHO Women's Health and Domestic Violence against Women Questionnaire will be used, which assesses emotional, sexual, and physical violence by intimate partners and has demonstrated good internal consistency ranging from 0.66 to 0.81.
Infant birthwight | At time of birth
  The infant's birth weight will be measured at the time of birth.
Gestational Age and Prematurity | At time of birth
  The gestational age of the infant at the time of birth will be measured. Premature infants are those whose gestational age is less than 37 weeks.
Infant diarrheal disease | Two weeks after infant's birth
  The occurrence of diarrheal disease among infants will be assessed during the first two weeks of the infant's life.
Weight-for-height | Up to 1.5 years after infant birth
  Wight and height will be measured as an outcome for the infant, with low weight-for-height being used to classify infants as wasting (more than two standard deviations below the mean).
Height-for-age | Up to 1.5 years after infant's birth
  Height and age of infants will be measured at the end of follow-up, and low height-for-age will be used to classify infants as stunted (more than two standard deviations below the mean).

CONTACTS AND LOCATIONS:
Overall Officials: Mary Kay Smith-Fawzi, ScD, Principal Investigator — Harvard Medical School (HMS and HSDM); Sylvia Kaaya, MD, PhD, Principal Investigator — Muhimbili University of Health and Allied Sciences
Locations (1):
- Dar es Salaam City Health Department, Dar es Salaam, Tanzania

REFERENCES:
- [Derived] Kaaya S, Siril H, Fawzi MCS, Aloyce Z, Araya R, Kaale A, Kasmani MN, Komba A, Minja A, Mwimba A, Ngakongwa F, Somba M, Sudfeld CR, Larson E. A peer-facilitated psychological group intervention for perinatal women living with HIV and depression in Tanzania-Healthy Options: A cluster-randomized controlled trial. PLoS Med. 2022 Dec 13;19(12):e1004112. doi: 10.1371/journal.pmed.1004112. eCollection 2022 Dec. PMID 36512631
- [Derived] Smith Fawzi MC, Siril H, Larson E, Aloyce Z, Araya R, Kaale A, Kamala J, Kasmani MN, Komba A, Minja A, Mwimba A, Ngakongwa F, Somba M, Sudfeld CR, Kaaya SF. Healthy Options: study protocol and baseline characteristics for a cluster randomized controlled trial of group psychotherapy for perinatal women living with HIV and depression in Tanzania. BMC Public Health. 2020 Jan 20;20(1):80. doi: 10.1186/s12889-019-7907-6. PMID 31959151